CLINICAL TRIAL: NCT05902923
Title: A Prospective PMCF Study Investigating the Safety and Clinical Performance of the Oceanus 18 and Oceanus 35 Balloon Dilatation Catheters, the Luminor 18 and Luminor 35 Drug Coated Balloons, the Restorer Peripheral Stent System, the iVolution Pro Peripheral Self-Expanding Stent System, the iCover Covered Peripheral Stent System and the Sergeant Peripheral Support Catheter for Endovascular Interventions.
Brief Title: Investigating the Safety and Clinical Performance of Eight iVascular Devices for Endovascular Intervention in Renal, Iliac or Femoral Arteries
Status: Recruiting | Type: Observational
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: FCRE-220209
Record Dates: First submitted 2022-03-28; First posted 2023-06-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention: All patients in the study will undergo same procedure. The implanted devices can be one of more of the study devices.
  Interventions: Procedure: endovascular intervention

INTERVENTIONS:
Procedure: endovascular intervention — endovascular intervention

SUMMARY:
The rationale of this study is to confirm and support the clinical safety and performance of any of these products in a real-world population of 209 patients who underwent an endovascular intervention within standard-of-care of the iliacofemoral artery and renal artery, using at least one of the investigational products from iVascular.

ELIGIBILITY:
Inclusion Criteria:

* Corresponding to the CE-mark indications/contra-indications and according to the IFU of the device.
* Patient is >18 years old.
* Patient understands the nature of the procedure and provides written informed consent prior to enrollment in the study.
* Target lesion(s) is/are located in renal, iliac or femoral arteries.
* Patient is eligible for treatment with the Oceanus 18 Balloon Dilatation Catheter and/or the Oceanus 35 Balloon Dilatation Catheter and/or the Luminor 18 Drug Coated Balloon and/or the Luminor 35 Drug Coated Balloon and/or the Restorer Peripheral Stent System and/or the iVolution pro Peripheral Self-Expanding Stent System and/or the iCover Covered Peripheral Stent System and/or the Sergeant Peripheral Support Catheter as described in IFU for each device.

Exclusion Criteria:

* Anatomy or size of vessels that will not allow appropriate usage of the investigational devices, following IFU of the investigational devices.
* Known contraindication and/or allergy to (a component of) an investigational device.
* Pregnant women and women with childbearing potential not taking adequate contraceptives or currently breastfeeding.
* Life expectancy of less than 12 months.
* Any planned surgical intervention/procedure within 30 days after the study procedure.
* Any patient considered to be hemodynamically unstable at onset of the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient who is eligible for treatment with any of the following devices, can be considered to be included in the study:
  the Oceanus 18 Balloon Dilatation Catheter and/or the Oceanus 35 Balloon Dilatation Catheter and/or the Luminor 18 Drug Coated Balloon and/or the Luminor 35 Drug Coated Balloon and/or the Restorer Peripheral Stent System and/or the iVolution pro Peripheral Self-Expanding Stent System and/or the iCover Covered Peripheral Stent System and/or the Sergeant Peripheral Support Catheter
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Freedeom from SAEs and SADEs (Primary Safety Endpoint) | during procedure and up to 2 years after procedure
  Freedeom from SAEs and SADEs
Technical success rate (Primary Efficacy Endpoint) | during procedure
  Technical success rate defined as ability to cross, introduce and deploy devices based on quantitative scaling by investigators

SECONDARY OUTCOMES:
General physician appraisal of the devices by means of rating scale | during procedure
  General physician appraisal of the devices will be explored based on: 1. Simplicity of handling, 2. Pushability, 3. Trackability, 4. Crossability and 5. Profile
General physician appraisal of the devices by means of rating scale for the Luminor 18, Luminor 35, Oceanus 18 and Oceanus 35 | during procedure
  Physician appraisal for the Luminor 18, Luminor 35, Oceanus 18 and Oceanus 35 will be explored based on: 1. Deflation time, 2. Balloon Compliance, 3. Visibility and 4. Balloon refolding
General physician appraisal of the devices by means of rating scale for the Restorer, iVolution pro, iCover | during procedure
  Physician appraisal for the Restorer, iVolution pro, iCover be explored based on: 1. Recoil, 2. Radial force, 3. Ease to canalize the lesion, 4. Stent coverage, 5. Stent graft recrossing and 6. Balloon refusal
General physician appraisal of the devices by means of rating scale for the Sergeant | during procedure
  And physician appraisal for the Sergeant will be explored based on: 1. Trackability over the guide wire, 2. Absence of kinking behaviour, 3. Injection Capacity, 4. Ease of changing guide wires and 5. Ease to canalize the lesion
Explorative endpoint | up to 2 years after procedure
  Freedom from SAEs and SADEs; Freedom from Target Lesion Revascularization

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH Henri Duffaut, Avignon
  - Clinique Synergia Ventoux, Carpentras
  - Polyclinique Inkermann, Niort
  - L'Hôpital Privé Des Côtes D'Armor, Plérin
  - Hôpital d'instruction des Armées Sainte Anne, Toulon
  - Hôpital Privé Toulon Hyeres St. Jean, Toulon